CLINICAL TRIAL: NCT03104270
Title: A Phase 2 Trial of the Efficacy and Safety of Elotuzumab in Combination With Pomalidomide, Carfilzomib and Dexamethasone Among High Risk Relapsed/ Refractory Multiple Myeloma Patients
Brief Title: Combination Study for High Risk Multiple Myeloma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by Funding Sponsor due to low enrollment.
Sponsor: Oncotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA204-187
Record Dates: First submitted 2017-02-27; First posted 2017-04-07 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma
Keywords: Elotuzumab, Multiple Myeloma, Phase 2
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; pomalidomide; carfilzomib; Dexamethasone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elo Pom Car and Dex (Experimental): Drug dosing and administration:
  All drugs are administered on a 28-day cycle.
  Elotuzumab: 10 mg/kg IV on Days 1,8,15 and 22 Cycles 1 and 2. 20 mg/kg on Day 1 of Cycles 3 and beyond.
  Pomalidomide: 3 mg PO on days 1-21
  Carfilzomib: 20 mg/m2 IV on days 1 of cycle 1. 56 mg/m2 IV on days 8 and 15 of cycle 1 and Days 1, 8 and 15 of the remaining seven cycles.
  Dexamethasone: On days 1,8,15,22 of Cycle 1-2 and day 1 of Cycle 3 and every day 1 thereafter, pre-treatment with 28 mg PO 3-24 hours prior to the start of ELO. On days 8,15,22 of Cycle 3 and beyond, 40mg of DEX PO or IV. On Day 8 and 15 of Cycle 3 and beyond, pre-treatment with DEX 40mg PO or IV at least 30 min and no more than 4 hours prior to the start of CFZ.
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab IV at 10mg/kg Elotuzumab IV at 20mg/kg
  Other Names: BMS-901608
Drug: Pomalidomide — Pomalidomide PO at 3mg
  Other Names: CC-4047, Pomalyst
Drug: Carfilzomib — Carfilzomib 20mg/m2 IV Carfilzomib 56mg/m2 IV
  Other Names: Kyprolis
Drug: Dexamethasone — Dexamethasone 28mg PO Dexamethasone 40mg PO or IV Dexamethasone 8mg IV
  Other Names: Steroid

SUMMARY:
Despite the recent introduction of novel anti-multiple myeloma (MM) agents, high risk MM remains with poor prognosis and a therapeutic challenge. Elotuzumab (ELO) is a humanized monoclonal antibody that recognizes CS1/CD139, a molecule highly expressed in MM cells. The ELO (10 mg/kg), lenalidomide (LEN) and dexamethasone (DEX) combination achieves high overall response rates (ORR) and long progression-free survival (PFS) for patients with relapsed/refractory disease (RR) MM and those with impaired renal function. However, its efficacy for MM patients with high risk characteristics is still unknown. Pomalidomide (POM) is a recently approved immunomodulatory agent (IMiD) that produces response rates for high-risk RRMM patients when used in combination with DEX and other agents, including the proteasome inhibitor (PI) bortezomib (BTZ). POM has also demonstrated activity for LEN refractory patients. Carfilzomib (CFZ) is a potent second generation PI that has shown to be efficacious for IMiD and BTZ refractory patients as well as high risk patients carrying cytogenetic abnormalities. In this study, we propose to evaluate efficacy and safety of ELO in combination with POM, DEX and CFZ for high-risk RRMM patients.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open label, nonrandomized study with six patients safety lead-in cohort to evaluate efficacy and safety of elotuzumab in combination with pomalidomide, carfilzomib and dexamethasone among high risk relapsed and refractory multiple myeloma patients.

This study will enroll previously treated patients that currently show evidence of progressive disease and have been diagnosed with high risk multiple myeloma. Thirty-nine patients will be enrolled in the study.

First, six patients will be enrolled and used as a lead-in cohort for the safety evaluation and MTD re-determination (if necessary). The results of the safety lead-in cohort will be evaluated after the 6th patient has completed one full cycle of treatment. Recruitment of patients will be withheld during safety data analysis. Enrollment of the remaining 33 patients will be contingent upon safety committee's decision.

The study consists of: 1) a screening period; 2) up to eight 28-day treatment cycles; 3) a final assessment to occur 28 days after the end of the last treatment cycle; and 4) a follow-up period.

All drugs will be administered on a 28-day cycle schedule throughout the study. Subjects eligible for this study will receive treatment with study drug for a maximum of eight 28-day treatment cycles. Subjects are to be treated for 8 cycles of therapy without demonstrating PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adults (age ≥ 18 years at the time of signing the informed consent document) and must meet all of the following inclusion criteria to be enrolled in the study:

  1. ECOG/Zubrod performance status of 0-2 at study entry
  2. Has a diagnosis of high-risk MM by showing any of the following a-f criteria: :

     1. Presence of conventional cytogenetic markers such as deletion of 17p-p53, translocations involving t(14;16) and t(14;20)
     2. Plasma cell leukemia (PCL) (> 2.0 × 109/L circulating plasma cells by standard differential)
     3. Extramedullary MM
     4. Doubling in levels of a MM markers in the past 3 months such as any of the following criteria alone or in combination: i) Serum M-protein ≥ 1.0 g/dL, or ii) Urine M-protein ≥ 400 mg/24 hours, or iii) Only in patients who do not meet i or ii, then use serum free light chain (SFLC) > 200 mg/L (involved light chain) and an abnormal kappa/lambda ratio
     5. Refractoriness to their most recent lenalidomide-containing regimen and proteasome inhibitor-containing regimen.
     6. Renal failure related to MM with creatinine clearance (CrCl) >15 mL/min but <30 mL/min as calculated by Cockcroft-Gault equation (Appendix 14.8).
  3. Has previously received more than two lines of therapy including a lenalidomide-containing regimen and proteasome inhibitor-containing regimen.
  4. Currently demonstrating progressive disease
  5. Life expectancy greater than 3 months
  6. Laboratory test results within these ranges at Screening and confirmed at enrollment prior to drug dosing on Cycle 1 Day 1:

     * ANC ≥ 1.5 x 109/L; if the bone marrow is extensively infiltrated ( ≥ 70% plasma cells) then ≥ 1.0 x 109/L
     * Platelet count ≥ 75 x 109/L; if the bone marrow is extensively infiltrated ( ≥ 70% plasma cells) then ≥ 50 x 109/L
     * Hemoglobin ≥ 8 g/dL
  7. Women of childbearing potential (WOCBP†) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 10-14 days prior to and again within 24 hours of starting study drug regimen

     † A WOCBP (women of childbearing potential) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle) for a total of 120 days post-treatment completion. Subject must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts taking study drugs. WOCBP must also agree to ongoing pregnancy testing. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Section 10.3.5.2, Appendix 4 and Appendix 5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of the study drug plus 90 days (duration of sperm turnover) for a total of 154 days post-treatment completion. Men must agree to use a latex condom during sexual contact with a WOCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Section 10.3.5, Appendix 4 and Appendix 5
  8. Able to take aspirin (acetylsalicylic acid, ASA) at 81 or 325 mg/daily as prophylactic anticoagulation (subjects intolerant to ASA may use warfarin or low molecular weight heparin)
  9. Written informed consent in accordance with federal, local, and institutional guidelines
  10. Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

  1. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) 19
  2. Waldenström's macroglobulinemia
  3. Received the following prior therapy:

     1. Elotuzumab
     2. Chemotherapy within 3 weeks of study drugs (6 weeks for nitrosourea, melphalan or monoclonal antibodies)
     3. Corticosteroids (>10 mg/daily prednisone or equivalent) within 3 weeks of study drugs
     4. Immunomodulatory therapy within one week before study drugs
     5. Antibody therapy within 3 weeks before study drugs
     6. Extensive radiation therapy (total maximum radiation doses of 50Gy to any individual site or 30Gy for the disseminated MM of bone) within 3 weeks before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
     7. Cytotoxic chemotherapy with approved or investigational anticancer therapeutics within 3 weeks prior to first dose
     8. Use of any other experimental drug or therapy within 3 weeks of study drugs
  4. Received the following transplant therapies:

     1. Less than 12 weeks from auto transplant
     2. Less than 16 weeks from allo transplant
     3. Less than 4 weeks since any plasmapheresis
  5. Major surgery within 4 weeks prior to first dose
  6. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

     1. Myocardial infarction within last 6 months prior to enrollment
     2. Active congestive heart failure (New York Heart Association (NYHA) Class III or IV) heart failure
     3. Uncontrolled angina and/or hypertension
     4. Clinically significant pericardial disease
     5. Severe uncontrolled ventricular arrhythmias
     6. Echocardiogram or MUGA evidence of LVEF below institutional normal within 28 days prior to enrollment
     7. Electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
  7. Known or suspected amyloidosis
  8. Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin
  9. Acute active infection requiring systemic antibiotics, antiviral), or antifungal agents
  10. Known positivity for human immunodeficiency virus (HIV)
  11. Known active hepatitis A,B or C virus infection
  12. Known active tuberculosis (TB) including subjects with latent TB or with the risk factor for activation of latent TB.
  13. Patients with known cirrhosis
  14. Secondary non-hematologic malignancy within the past 3 years, except:

      1. Adequately treated basal cell or squamous cell skin cancer
      2. Carcinoma in situ of the cervix
      3. Prostate cancer < Gleason score 6 or less with stable prostate-specific antigen (PSA) levels over 12 months
      4. Breast carcinoma in situ with full surgical resection
      5. Treated medullary or papillary thyroid cancer
  15. Patients with myelodysplastic syndrome
  16. Prior cardio vascular accident (CVA) with persistent neurological deficit
  17. Significant neuropathy (Grades 3 to 4) within 14 days prior to first dose
  18. Peripheral neuropathy with pain ≥ G2 within 14 days prior to first dose
  19. Women who are pregnant and/or breast feeding
  20. Known hypersensitivity to dexamethasone
  21. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
  22. Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide
  23. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
  24. Hypersensitivity to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs.
  25. Ongoing graft-versus-host disease.
  26. Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment.
  27. Uncontrolled diabetes within 2 weeks prior to enrollment.
  28. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 34 Months
  Occurrence of adverse events throughout the study, graded via Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 criteria (If necessary re-define MTD via the number of dose-limiting toxicities (DLTs) per dose level, of elotuzumab in combination with pomalidomide, carfilzomib and dexamethasone for high risk RRMM patients (based on six patients lead-in cohort if necessary).
Overall Rate of Response (Efficacy) | 34 Months
  Efficacy of treatment will be assessed by the Overall response rate (ORR) [ORR=complete response (CR†) + very good partial response (VGPR) + partial response (PR)] Clinical benefit rate (CBR) [CBR=CR† + VGPR + PR + minor response (MR)].

SECONDARY OUTCOMES:
PFS | 34 Months
  Progression-free survival (PFS): time from initiation of therapy to progressive disease or death from any cause, whichever comes first
DOR | 34 Months
  Duration of response (DOR): time from the first response (> PR) to progressive disease
OS | 34 Months
  Overall survival (OS): time from initiation of therapy to death from any cause or last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (6):
- United States (6):
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - Robert A. Moss, MD, FACP, Inc, Fountain Valley, California
  - Pacific Cancer Care, Monterey, California
  - James Berenson, MD, Inc, West Hollywood, California
  - Millennium Oncology Research Clinic, Pembroke Pines, Florida
  - Regional Cancer Care Associates MD LLC, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yashar D, Spektor TM, Martinez D, Ghermezi M, Swift RA, Eades B, Schwartz G, Eshaghian S, Lim S, Vescio R, Berenson JR. A phase 2 trial of the efficacy and safety of elotuzumab in combination with pomalidomide, carfilzomib and dexamethasone for high-risk relapsed/refractory multiple myeloma. Leuk Lymphoma. 2022 Apr;63(4):975-983. doi: 10.1080/10428194.2021.2005044. Epub 2021 Nov 24. PMID 34818965